CLINICAL TRIAL: NCT03899038
Title: Minimum Effective Dose of 0.5% Bupivacaine for Ultrasound-guided Spinal Anesthesia Using Taylor's Approach
Acronym: MEDBST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Vice Director, Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: US-Spinal
Record Dates: First submitted 2019-03-27; First posted 2019-04-02 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Lower Limb Surgery
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deceasing (Experimental): Spinal anesthesia with decreasing dose. Real-time ultrasound-guided spinal anesthesia Using Taylor's approach.
  Interventions: Procedure: spinal anesthesia
- Similar (Active Comparator): Spinal anesthesia with similar dose. Real-time ultrasound-guided spinal anesthesia Using Taylor's approach.
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — Patients will receive real-time ultrasound guided spinal anesthesia using Taylor's approach. Various doses of bupivacaine 0.5% (Bupivacaine hydrochloride injection, Harvest Pharmaceutical CO., LTD., Shanghai, China) will be administered.

SUMMARY:
This study aims to determine the minimum effective dose of bupivacaine 0.5% in 90% of patients undergoing lower limb surgery with ultrasound-guided spinal anesthesia using Taylor's approach. A biased coin design up-and-down sequential method is applied. The initial dose is 15 mg of bupivacaine 0.5%. After 45 successful spinal anesthesia, the ED90 of bupivacaine 0.5% will be calculated.

DETAILED DESCRIPTION:
The minimum effective dose of local anesthetics for spinal anesthesia using Taylor's approach is not known. This study aims to determine the minimum effective dose of bupivacaine 0.5% using a biased coin design up-and-down sequential method. Patients will receive real-time ultrasound guided spinal anesthesia using Taylor's approach. The initial dose is chosen as 15 mg on the basis of clinical experience. Subsequently, if a patient has an inadequate block, the bupivacaine dose is increased by 2 mg in the next subject. If a patient has a successful block, the next subject is randomized to receive either a lower dose (with a decrement of 2 mg), with a probability of b = 0.11, or the same dose, with a probability of 1 - b = 0.89. Forty five successful blocks will be accomplished. MED90 will be calculated by isotonic regression.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical statusⅠ- Ⅲ
* Lower limb surgery, expected operation time within 2 hours

Exclusion Criteria:

* Patient refusal
* American Society of Anesthesiologists physical status IV/V
* Peripheral neuropathy
* skin infection at the site of injection
* allergy to bupivacaine or lidocaine
* BMI > 35 kg/m2
* coagulation disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The minimum effective dose of bupivacaine in spinal anesthesia using Taylor's approach | up to 6 months
  The minimum effective dose of bupivacaine in spinal anesthesia using Taylor's approach is based on 45 successful spinal anesthesia performed in patients undergoing lower limb surgery.

SECONDARY OUTCOMES:
the upper level of the sensory block 25 min after bupivacaine injection | 25 min
  the upper level of the sensory block 25 min after bupivacaine injection
the incidence of hypotension | during anethesia and operation
  the incidence of hypotension
the duration of sensory spinal anaesthesia for the lower extremity | up to 3 days postoperation
  the duration of sensory spinal anaesthesia for the lower extremity
postoperative neurological complications | up to 3 months postoperation
  postoperative neurological complications

CONTACTS AND LOCATIONS:
Overall Officials: Mujun Chang, MD, Study Director — Tongji Hospital,Wuhan
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No